CLINICAL TRIAL: NCT05064228
Title: Mobile Health Intervention to Increase Substance-Free Reward During Alcohol Treatment
Brief Title: Mobile Rewarding Activity Centered Treatment
Acronym: mReACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Lidia Meshesha, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AWD00000705
Record Dates: First submitted 2021-09-03; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: ecological momentary assessment; ecological momentary intervention; Alcohol Use Disorder Treatment; Adjunctive intervention
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the m-ReACT intervention condition or an active control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- m-ReACT app condition (Experimental): Participants will download the m-ReACT app on their mobile phones and will be asked to engage with the app for a period of 12 weeks.
  Interventions: Behavioral: Mobile Rewarding Activity Centered Treatment (m-ReACT)
- Brief Advice (Active Comparator): Participants will be given a one time brief informational session on the importance of engaging in substance-free activity while in AUD treatment.
  Interventions: Behavioral: Mobile Rewarding Activity Centered Treatment (m-ReACT)

INTERVENTIONS:
Behavioral: Mobile Rewarding Activity Centered Treatment (m-ReACT) — Participants will utilize m-ReACT for 12-weeks, reporting daily on substance-free activity engagement and enjoyment (EMA). m-ReACT will utilize these EMA reports to generate brief, automated, and personalized feedback about enjoyed categories of substance-free activities as well as make suggestions for increasing engagement in those rewarding, goal-oriented substance-free activities, and provide personalized suggestions of activities of interest.

SUMMARY:
Alcohol Use Disorder (AUD) is a highly prevalent and significant public health problem. Behavioral treatments based in the principles of social learning theory and cognitive behavior therapy have been developed and tested for AUD, yet effect sizes are relatively small and rates of relapse following treatment are high. Theoretically informed adjunctive interventions may help to enhance the effects of extant AUD treatments. In particular, evidence suggests that environments lacking in substance-free (SF) activities contribute to the development and maintenance of AUD and that the availability of rewarding SF activities may serve as viable alternatives to compete with alcohol use. Building on the advantages of accessibility and low-cost option afforded by the use of mobile technology, this proposal outlines a well-integrated research and training plan to investigate a mobile health intervention to increase engagement in rewarding SF activities among patients in AUD treatment. This proposed research aims to develop and evaluate a mobile phone ecological momentary assessment plus ecological momentary intervention (EMA+EMI; entitled: mobile - Rewarding Activity Centered Treatment (m-ReACT)) app to augment existing AUD treatment. The m-ReACT app will monitor self-reported rewarding SF activity engagement in real-time and deliver personalized feedback that encourages participants to engage in highly rewarding activities that are goal-oriented and support positive treatment outcomes. This proposed intervention will be developed in two phases. Phase 1 will develop the m-ReACT app and Phase 2 will evaluate its efficacy in randomized control pilot trial with a sample of 50 AUD patients who have recently initiated outpatient AUD treatment. Participants in the pilot RCT will be randomly assigned to either the m-ReACT condition or an active control condition. It is hypothesized that m-ReACT will result in increased rates of percent days of alcohol abstinence and increased reinforcement from SF activities.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is strongly linked with deficits in alcohol-free alternative rewards. Individuals with AUD have limited sources of substance-free (SF) natural rewards. Increasing SF rewards in the context of treatment is of immediate public health relevance as it has the potential to improve AUD treatment outcomes. Yet, this is not a focus of standard outpatient treatment. Prior studies demonstrate that interventions focused on SF alternatives in addition to standard treatment improve outcomes above and beyond standard treatment alone. However, these efficacious treatments can be difficult to implement and sustain within a real-world AUD treatment facility. Therefore, it is essential to enhance the approach used in these studies to meet the needs of patients and treatment facilities alike. Novel methodologies that are cost effective, technologically enhanced, and less time intensive are needed to better incorporate this intervention within a treatment setting. The proposed study would make use of mobile technology to aid patients engage in alternative behaviors, who otherwise may have limited access to activities other than drinking, and thereby potentially help reduce risk of relapse.

This research proposal aims to develop and evaluate an ecological momentary intervention (EMI) supported by an ecological momentary assessment (EMA) aimed at increasing reinforcement from substance-free activities among AUD patients in order to improve treatment outcomes. Towards this end, this research will be conducted in two phases. Phase 1 will entail an iterative process of EMA plus EMI development of a smartphone app, called mobile-Rewarding Activity Centered Treatment (m-ReACT), designed to collect real-time data on substance-free activity engagement and obtained reward. The data will then be provided back to the individuals to encourage engagement in activities that were most rewarding.

Upon app successful app development, this study will implement phase 2. Phase 2 will consist of a pilot RCT (N=50) to evaluate m-ReACT as an adjunctive intervention for AUD treatment-seekers compared to a brief advice (BA) session on engaging in SF pleasant activities. Participants will be randomized to either an in-person informational session consisting of BA on the importance of engaging in SF rewarding activities or brief in-person app orientation session that will collect daily reporting of substance free activity engagement and enjoyment and provide personalized feedback on level of substance free activity engagement and enjoyment with encouragement to continue engagement. Feasibility and acceptability of m-ReACT will be assessed with self-report measures, qualitative end-of treatment interviews, and examination of app usage from the app metadata. Follow-up assessments will be conducted at 3 (end of treatment) and 6-months to evaluate for drinking related outcomes and SF reinforcement.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 65 years of age
2. primary DMS-5 diagnosis of AUD
3. currently enrolled in outpatient treatment of AUD
4. Own a smarphone

Exclusion Criteria:

1. enrolled to attend higher level of care (i.e., inpatient or residential treatment) after discharge from current outpatient treatment program
2. a history of psychotic disorder or current psychotic symptoms
3. current suicidal or homicidal ideation
4. moderate or severe DSM-5 substance use disorders other than alcohol or nicotine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow-Back - Change in drinking over time | This will be assessed at baseline, 3months, and 6months post baseline
  The 90-day timeline follow-back will be used to asses change over time in percent days abstinent from alcohol

SECONDARY OUTCOMES:
Reward Probability Index - Change over time | This will be assessed at baseline, 3months, and 6months post baseline
  The study will assess change in for RPI substance free reinforcement
Temporal Experience of Pleasure Scale - Change over time | This will be assessed at baseline, 3months, and 6months post baseline
  Assess change over time in experience of pleasure as a measure of substance free reinforcement
SF Pleasant Image Ratings - Change over time | This will be assessed at baseline, 3months, and 6months post baseline
  Assess change over time in objective pleasant image ratings as a measure of substance free reinforcement

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be shared with NIH Data Archive
Time Frame: As data gets collected starting December 2023 throughout end of data collection with no planned end date
Access Criteria: Individuals or organizations with access to NIH Data Archive